CLINICAL TRIAL: NCT00062985
Title: Obesity Treatment in a Managed Care Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OBMANC (completed); R01DK053826 (NIH)
Record Dates: First submitted 2003-06-18; First posted 2003-06-19 (Estimated); Last update posted 2017-10-24 (Actual); Status verified 2017-10

CONDITIONS: Obesity; Weight Loss
Keywords: obesity treatment; weight management; managed care
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention)
- Mail-based weight loss intervention (Experimental)
  Interventions: Behavioral: Mail-based weight loss intervention
- Telephone-based weight loss intervention (Experimental)
  Interventions: Behavioral: Phone-based weight loss intervention

INTERVENTIONS:
Behavioral: Mail-based weight loss intervention
  Arms: Mail-based weight loss intervention
Behavioral: Phone-based weight loss intervention
  Arms: Telephone-based weight loss intervention

SUMMARY:
The aim of the present study is to evaluate the effectiveness of two different delivery formats for weight management in a managed care setting. Mail-based weight counseling and phone-based weight counseling will be compared to each other and a control condition. Primary outcomes are participation rates in programs, weight change, and cost.

ELIGIBILITY:
* at least 18 years of age
* BMI ≥ 27.8 kg/m2 for men
* BMI ≥ 27.3 kg/m2 for non-pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1801 (Actual)
Dates: Start 1999-03 (Actual); Primary Completion 2003-10 (Actual); Study Completion 2005-02 (Actual)

PRIMARY OUTCOMES:
Change in body weight | 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Robert W. Jeffery, PhD, Principal Investigator — University of Minnesota, Division of Epidemiology
Locations (1):
- University of Minnesota, Division of Epidemiology, Minneapolis, Minnesota, United States

REFERENCES:
- [Result] Jeffery RW, Sherwood NE, Brelje K, Pronk NP, Boyle R, Boucher JL, Hase K. Mail and phone interventions for weight loss in a managed-care setting: Weigh-To-Be one-year outcomes. Int J Obes Relat Metab Disord. 2003 Dec;27(12):1584-92. doi: 10.1038/sj.ijo.0802473. PMID 14517547